CLINICAL TRIAL: NCT05825924
Title: Randomized, Two Arm Parallel, Clinical Trial to Compare Effectiveness of Different Tobacco Harm Reduction Products in General Adult Population in Low Middle Income Countries
Brief Title: Effectiveness of Different THR Products in Adult Population
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Foundation for a Smoke Free World INC (Other)
Responsible Party: Principal Investigator, Dr. Madeeha Malik, Principal Investigator, Foundation for a Smoke Free World INC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W3-030
Record Dates: First submitted 2023-03-14; First posted 2023-04-24 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; tobacco harm reduction; E Cigarettes; LMIC
MeSH Terms: conditions — Smoking Cessation; Vaping | interventions — Tobacco Use Cessation Devices; Transdermal Patch

STUDY DESIGN:
Intervention Model Description: Participants who are eligible and consent to take part will be randomized (1:1 ratio) to receive products accordingly: A total of 258 participants will be enrolled (129 in each arm) and randomized to Study Arm A: 18 mg nicotine e-cigarettes (ad libitum use) for 12 weeks after the nominated quit date; and Study Arm B: 21 mg nicotine patches (one daily) for 12 weeks after the nominated quit date. The duration of counseling will be at least 30 minutes at site. The duration of counseling through telephone will be at least 10 minutes. Participants will be scheduled for a screening visit and a baseline (BL) visit at the trial site. The participants will be scheduled for eight study visits in total, including five treatment sessions and three follow-up visits, using both face to face interaction at trial site as well as follow up on telephone. Eight study visits are planned at weeks 1, 2, 4, 8, 12, 18, 24, and 52.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Study Arm A: Electronic Cigarettes (18mg/ml) (Active Comparator): Participants randomized to study arm A will be provided a free e-cigarette and sufficient nicotine cartridges (18 mg/ml) supply to last till next in person visit. Participants will be instructed to use the device ad libitum one week before their quit day to familiarize themselves with its operation and on their designated quit day will stop smoking tobacco cigarettes and instead use the e-cigarette exclusively for the next 12 weeks. Smokers often take 10 to 15 puffs over the course of 5 to 8 minutes, repeating this pattern with each cigarette. On the other hand, users of EC may periodically use it throughout the day, and they may or may not take their puffs like those of traditional cigarettes
  Interventions: Device: E-Cigarette
- Study Arm B: 21 mg nicotine patches (Active Comparator): Participants randomized to study arm B will be provided 21 mg nicotine patches supply to last till next in person visit. Participants will use the nicotine patch daily for one week before their quit day to familiarize themselves with its use. On their designated quit day they will stop smoking and use nicotine patches daily for the next 12 weeks. Usually a full-strength patch (15-22 mg of nicotine) daily for four weeks is suggested for use in majority of the smokers, followed by a lower strength patch (5-14 mg of nicotine) for an additional four weeks, depending on their body size and smoking habits
  Interventions: Drug: Nicotine patch

INTERVENTIONS:
Device: E-Cigarette — E-cigarettes have been designed to resemble tobacco cigarettes. They include an aerosol generator, sensor, battery and storage area for liquid. They are either disposable or rechargeable. According to a study, e-cigarettes can deliver an average of 1.3 mg (range 0.4 to 2.6 mg) of nicotine from 15 puffs. Average Cmax after e-cigarette use is recorded as 8.4 ng/mL and Tmax achieved between 2 to 5 minutes
  Arms: Study Arm A: Electronic Cigarettes (18mg/ml)
Drug: Nicotine patch — The nicotine patches are applied on the skin and nicotine is delivered at a steady rate. After administration, the peak blood levels are achieved within 6-10 hours. The levels remain constant, reducing by 25-40% with use of patches once daily. The patch is typically administered every 24 hours for no longer than 12 weeks. The dose of the patches is often determined by daily cigarette consumption and level of addiction.
  Other Names: Patch
  Arms: Study Arm B: 21 mg nicotine patches

SUMMARY:
The study is a two-arm, parallel randomized controlled trial (RCT) with a treatment period of 12 weeks, and long-term follow-up at 52 weeks which plans to enroll 258 smokers from general adult population. Participants who meet the eligibility criteria and give their informed consent will be randomized (1:1) to one of two treatment arms: (1) E-cigarettes (18mg/ml) with individual counselling (2) Nicotine patches (21mg) with individual counselling. Eligible participants must be at least of legal age allowed for smoking in the country, of either gender, regular smokers (minimum 10 cigarettes/day for at least a year) and interested to stop smoking. Participants will be scheduled for a screening visit and a baseline (BL) visit at the trial site. The participants will be scheduled for eight study visits in total, including five treatment sessions and three follow-up visits, using both face to face interaction at trial site as well as follow up on telephone. Eight study visits are planned at weeks 1, 2, 4, 8, 12, 18, 24, and 52. Exhaled carbon monoxide assessment will be used at the trial site to quantify biochemically validated smoking abstinence. All secondary outcomes and self-reported usage of nicotine patches, EC and cigarettes will be monitored throughout the study.

DETAILED DESCRIPTION:
This is a two-arm, parallel randomized controlled trial with a 12 weeks treatment duration and long-term 52 weeks follow-up. Outpatient, and walk-in clinics, and advertising will be used to recruit participants from the general population. Individual counselling regarding smoking cessation will be provided to the participants using EC as well as nicotine patches. Participants included must be at least of legal age allowed for smoking in the country, of either gender, regular smokers (minimum 10 cigarettes/day for at least a year) and interested to stop smoking. Participants will be scheduled for a screening visit and a baseline (BL) visit at the trial site. The participants will be scheduled for eight study visits in total, including five treatment sessions and three follow-up visits, using both face to face interaction at trial site as well as follow up on telephone. Eight study visits are planned at weeks 1, 2, 4, 8, 12, 18, 24, and 52. Exhaled carbon monoxide assessment will be used at the trial site to quantify biochemically validated smoking abstinence (exhaled carbon monoxide levels above ten ppm regarded as indicator of current smoking). All secondary outcomes and self-reported usage of nicotine patches, EC and cigarettes will be monitored throughout the study. Information about self-reported smoking, usage of EC and nicotine patches, use of other smoking cessation therapy and side effects will be gathered at all follow-up calls and visits.

ELIGIBILITY:
Inclusion Criteria:

* Both genders of legal age allowed for smoking as per country law
* Smoked at least 10 cigarettes a day for the past one year
* Exhaled breath CO (eCO) level > 10 ppm
* Wish to quit smoking
* Able to conform with all study procedures
* Have a mobile phone
* Expected to be available for follow up will be enrolled as study participants

Exclusion Criteria:

* Pregnant and breastfeeding women
* Using other smoking cessation medications (including other forms of NRT other than patch, bupropion, clonidine, nortriptyline or varenicline)
* Having any contraindications to products such as cardiovascular history
* Suffering from a major illness with prognosis of less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Point-prevalence abstinence | 12 weeks
  Number of participants self-reported abstinence in the past week, with biochemical validation using exhaled CO measurements of ≤ 10 ppm.

SECONDARY OUTCOMES:
Seven-day point prevalence | 7 days for 12 weeks
  Number of Participants who self-report having smoked no cigarettes in the past 7 days
Use of tobacco combustible cigarettes | 12 weeks
  Number of cigarettes smoked per day assessed using self reported diaries
Perception of the product | 12 weeks
  Participant views on using e-cigarettes or patches as a smoking cessation aid using Modified Cigarette Evaluation Questionnaire. The mCEQ consist of 12 questions for rating using Likert scale which ranges from 1 (not at all) to 7 (extremely). The answers are combined to form five unique subscales each made up of 1-5 items which quantify (1) Satisfaction, (2) Psychological Reward, (3) Enjoyment of Respiratory Tract Sensations, (4) Craving and (5) Aversion. Difference scores can range from -6 to +6 with positive scores indicating higher dose cigarette produce greater intensity of a subjective effect.
Adverse events | 12 weeks
  Adverse events related to e cigarettes and nicotine patches evaluated using Naranjo Adverse Drug Reaction Probability Scale. Total scores range from -4 to +13 with higher scores indicating definite adverse drug reaction; the reaction is considered definite and adverse reaction is present if the score is 9 or higher, probable if 5 to 8, possible if 1 to 4, and doubtful if 0 or less.
Physical signs and symptoms associated with withdrawal | 52 weeks
  Physical sign and symptoms of withdrawal using Fagerstrom test for nicotine dependence. It contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence. In scoring the Fagerstrom Test for Nicotine Dependence, yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are computed to yield a total score of 0-10. The higher the total Fagerstrom score, the more intense is the participant's physical dependence on nicotine.

CONTACTS AND LOCATIONS:
Overall Officials: Madeeha Malik, PhD, Principal Investigator — Cyntax Health Projects PVT LTD
Locations (1):
- South East Hospital and Research Centre, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No